CLINICAL TRIAL: NCT07039734
Title: Assessment of Ovarian Reserve in Patients With Fragile X Premutation
Acronym: ROFRA
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP250753
Record Dates: First submitted 2025-05-14; First posted 2025-06-26 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: FMR1 Gene Premutation
Keywords: POI; ovarian reserve; fertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: collection of data from medical records — collection of data from medical records

SUMMARY:
Premature ovarian failure (POF) affects 1% of women under the age of 40 and is defined by the presence of a disorder of the cycle such as spaniomenorrhea or amenorrhea and an increase in FSH > 25 IU/l on two occasions a few weeks apart.

The prevalence of premature ovarian failure in women carrying the FMR1 gene premutation is estimated to be between 13 and 26%. Conversely, patients carrying premutations have been identified in 0.8 to 7.5% of women with sporadic POI and up to 13% of women with a familial form of POI.

The variability in penetrance seems to be due, among other things, to the increased probability of POI with the increased number of CGG repeats. This relationship is not linear; indeed, the risk appears to increase with the increase in the number of CGG triplets between 59 and 99, then the risk reaches a plateau or even decreases for women with more than 100 repeats. Patients with a full FMR1 mutation are not at a higher risk of POI than the general population.

The systematic evaluation of ovarian function and reserve in patients with FMR1 premutation and the monitoring of the latter over time is therefore a major element in the management of these women in order to be able to provide them with advice regarding their fertility or even to discuss ways of preserving their fertility. There are no longitudinal data on the evolution of ovarian reserve over time in pre-matured women, nor is there any determination of early predictive factors for its alteration.

We propose to retrospectively evaluate ovarian function and its evolution over time in pre-matured women seen in 2 reference centers (Paris, Lyon) based on questionnaires, blood tests and pelvic ultrasound.

DETAILED DESCRIPTION:
Premature ovarian failure (POF) affects 1% of women under the age of 40 and is defined by the presence of a disorder of the cycle such as spaniomenorrhea or amenorrhea and an increase in FSH > 25 IU/l on two occasions a few weeks apart.

The prevalence of premature ovarian failure in women carrying the FMR1 gene premutation is estimated to be between 13 and 26%. Conversely, patients carrying premutations have been identified in 0.8 to 7.5% of women with sporadic POI and up to 13% of women with a familial form of POI.

The variability in penetrance seems to be due, among other things, to the increased probability of POI with the increased number of CGG repeats. This relationship is not linear; indeed, the risk appears to increase with the increase in the number of CGG triplets between 59 and 99, then the risk reaches a plateau or even decreases for women with more than 100 repeats. Patients with a full FMR1 mutation are not at a higher risk of POI than the general population.

The systematic evaluation of ovarian function and reserve in patients with FMR1 premutation and the monitoring of the latter over time is therefore a major element in the management of these women in order to be able to provide them with advice regarding their fertility or even to discuss ways of preserving their fertility. There are no longitudinal data on the evolution of ovarian reserve over time in pre-matured women, nor is there any determination of early predictive factors for its alteration.

We propose to retrospectively evaluate ovarian function and its evolution over time in pre-matured women seen in 2 reference centers (Paris, Lyon) based on questionnaires, blood tests and pelvic ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* - Women aged 18 to 40 years old, carriers of FMR1 premutation, regardless of the number of CGG triplet repeats
* Informed patients who do not object to participating in the research- Patients who have been informed and do not object to participating in the research

Exclusion Criteria:

* - Gynecological history that may have impacted ovarian reserve: surgery, radiotherapy, chemotherapy or endometriosis
* Patients who are not affiliated with a social security scheme or who are not entitled to it
* Patients under legal protection, or under guardianship or trusteeship.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patient with FMR1 premutation followed in one of the two recruiting departments.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-07-04 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
characterize ovarian reserve in women diagnosed with FMR1 premutation | Day1
  AMH dosage

SECONDARY OUTCOMES:
Gonadotrophic axis at diagnosis and annually | at diagnosis and annually
Endovaginal pelvic ultrasound with counting of antral follicles at diagnosis and annually | at diagnosis and annually
Duration of menstrual cycles | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Endocrinologie et médecine de la reproduction Hôpital Pitié-Salpêtrière, Paris, France, France

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.